CLINICAL TRIAL: NCT06481813
Title: BREATHE Cohort : Prospective, Longitudinal Biocollection in Thoracic Oncology, Including Newly Diagnosed Lung Cancer Patients
Brief Title: Prospective, Longitudinal Biocollection in Thoracic Oncology, Including Newly Diagnosed Lung Cancer Patients
Acronym: BREATHE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC21_0541; 2024-A00509-38 (Other: ANSM (IDRCB))
Record Dates: First submitted 2024-05-23; First posted 2024-07-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Metastatic Lung Cancer
Keywords: Real-world cohort; Lung Cancer; Biobank
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This cohort will include 5 distinct patient populations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort A (Other): Patients are prospectively enrolled the day before their surgery for lung cancer, following selection based on tumor size assessed by the latest CT scan. The lesion size must be ≥ 20 mm (to prioritize anatomopathological analyses performed as part of care). If patients receive adjuvant treatment, blood samples will be collected on the day of treatment initiation and during follow-up. Patients receiving neoadjuvant treatment will be enrolled at the time of their first consultation with the medical oncologist.
  Patients in this cohort must meet the following criteria:
  - Stage I / II / IIIA-B localized NSCLC (non-small-cell lung cancer) eligible for surgery and adjuvant or neoadjuvant therapy (15-20% of NSCLC)
  Intervention : patients will be sampled from 2 x 8 mL blood tubes (EDTA tubes)
  Interventions: Other: Blood Sampling (2*8mL Tubes)
- Cohort B (Other): Patients are prospectively enrolled at the diagnosis of lung neoplasm, during the establishment of the therapeutic plan by the referring oncologist or pneumo-oncologist. Enrollment can also occur at the initiation of first-line treatment if it was not done at the time of the diagnostic consultation.
  Patients in this cohort must meet the following criteria:
  - metastatic NSCLC or SCLC (small-cell bronchial cancers), with drained or punctured pleural effusion and anatomopathological evidence of tumor cells
  Intervention, the following volumes of blood will be drawn at each visit :
  * 2*8ml (EDTA tubes)
  * 1*8mL PBMC (only for patients receiving immunotherapy, collected before the 1st course of treatment, before the 2nd course of treatment, and at relapse)
  * 1*6mL Paxgene (only for patients with lung cancer of non-epidermoid histology, collected at 1st treatment, 2nd treatment and relapse)
  Interventions: Other: Blood Sampling (2*8mL Tubes); Other: PBMC Sampling (1*8mL Tubes); Other: Paxgene Sampling
- Cohort C (Other): Cohort C patients are recruited in the same way as for cohort B.
  Patients in this cohort must meet the following criteria:
  * Metastatic NSCLC receiving systemic chemotherapy, immunotherapy and/or targeted therapy
  * Locally advanced stage III NSCLC treated with radio-chemotherapy +/- immunotherapy
  * Extra-thoracic SCLC treated with chemotherapy +/- immunotherapy
  * Intra-thoracic SCLC treated with radio-chemotherapy
  Intervention, the following volumes of blood will be drawn at each visit :
  * 2*8ml (EDTA tubes)
  * 1*8mL PBMC (only for patients receiving immunotherapy, collected before the 1st course of treatment, before the 2nd course of treatment, and at relapse)
  * 1*6mL Paxgene (only for patients with lung cancer of non-epidermoid histology, collected at 1st treatment, 2nd treatment and relapse)
  Interventions: Other: Blood Sampling (2*8mL Tubes); Other: PBMC Sampling (1*8mL Tubes); Other: Paxgene Sampling
- Cohort BMB (Other): Patients are enrolled preoperatively, at the diagnosis of metastatic lung cancer at the cerebral level. The patient signs consent preoperatively (consent provided by the neurosurgeon). Subsequently, they are prospectively followed as part of their management in medical oncology, postoperatively.
  Patients in this cohort must meet the following criteria:
  - Patient operated on for brain metastasis as part of care, and diagnosed with lung cancer.
  Intervention, the following volumes of blood will be drawn at each visit :
  * 2*8ml (EDTA tubes)
  * 1*8mL PBMC (only for patients receiving immunotherapy, collected before the 1st course of treatment, before the 2nd course of treatment, and at relapse)
  * 1*6mL Paxgene (only for patients with lung cancer of non-epidermoid histology, collected at 1st treatment, 2nd treatment and relapse)
  Interventions: Other: Blood Sampling (2*8mL Tubes); Other: PBMC Sampling (1*8mL Tubes); Other: Paxgene Sampling
- Healthy Controls : (Other): A population of healthy subjects will also be included. These healthy subjects will be either :
  * Companions of patients with lung cancer who have come to the oncology clinic for their loved ones.
  * Patients who have undergone atypical lung resection as part of their care for pneumothorax.
  Intervention : Healthy subject will be sampled from 2 x 8 mL blood tubes (EDTA tubes)
  In addition to blood samples from healthy subjects, healthy tissue remnants from atypical lung resections performed as part of care for pneumothorax management will be used to analyze the study objectives.
  A maximum of 30 healthy subjects are expected in this population.
  Interventions: Other: Blood Sampling (2*8mL Tubes)
- Ancillary study (Other): Patients included in the other arms of the cohort may also participate in the ancillary study if they meet the following conditions :
  Being carriers of metastatic KRAS G12C mutated NSCLC with a treatment plan involving sotorasib, adagrasib, or another KRAS inhibitor, either alone or in combination with another treatment.
  A target of 40 patients (among the 700 patients included in the cohort, excluding healthy subjects) is set for the ancillary study.
  Interventions: Procedure: Extended biopsies of tumor lesions

INTERVENTIONS:
Other: Blood Sampling (2*8mL Tubes) — Patients will be sampled from 2 x 8 mL blood tubes (EDTA tubes)
  Arms: Cohort A; Cohort B; Cohort BMB; Cohort C; Healthy Controls :
Other: PBMC Sampling (1*8mL Tubes) — Patients will be sampled from 1 x 8 mL PBMC
  Arms: Cohort B; Cohort BMB; Cohort C
Other: Paxgene Sampling — Patients will be sampled from 1 x 8 mL of blood with Paxgene Tube
  Arms: Cohort B; Cohort BMB; Cohort C
Procedure: Extended biopsies of tumor lesions — Regarding the ancillary study, as part of the care, patients are biopsied at diagnosis and during relapse(s). For metastatic patients with multiple sites, one site (the most accessible) is chosen and biopsied in interventional radiology or pulmonology.
  The material used is: 17-18G biopsy needle / Sampling chamber volume of 0.01 cm³ to 0.02 cm³.
  For a standard biopsy as part of the care, 3 samples are taken (total volume of 0.03 cm³ to 0.06 cm³). Inclusion in the ancillary study would add one sample using the same biopsy path, resulting in an additional volume of 0.01 cm³ to 0.02 cm³.
  In the case of a complex biopsy, no additional sampling related to the research will be performed.
  Arms: Ancillary study

SUMMARY:
In clinical trials, patients are selected according to strict eligibility criteria (inclusion and exclusion criteria). These criteria aim to ensure homogeneity within the trial population, but may omit patients with specific characteristics, comorbidities or co-medications. Indeed, patients of advanced age, with comorbidities or brain metastases, who are frequently encountered in clinical practice, are often excluded from clinical trials. Real-life data in oncology play a vital role in assessing the efficacy of therapies and therapeutic strategies, complementing data from controlled clinical trials. They make it possible to analyze a larger population and take into account multiple variables such as patient history, co-medications and comorbidities, but also to analyze efficacy and toxicity data in populations not represented in clinical trials. The establishment of a prospective cohort including various stages and histologies will make it possible to set up a platform of available data, including a maximum of data linked to the patient, his tumor and his treatments, collected longitudinally until the patient's death (or the end of the study).

In parallel with this cohort, the project aims to set up a longitudinal plasmatheque (from diagnosis to death, or at the end of the study), as well as a tumorotheque (samples systematically stored as part of care by the CHU tumorotheque, and for which patient consent allows their use in research depending on the material available) for patients with available tumor samples. This will enable the construction of ancillary projects to validate research hypotheses, for example concerning the identification of mechanisms of resistance to therapies.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Adult
* Patient newly diagnosed with NSCLC or CPC
* Cared for at Nantes University Hospital
* Affiliated or beneficiaries of a social security scheme or similar
* Treated with a systemic therapy including chemotherapy and/or immunotherapy and/or targeted therapy and/or therapy as part of a clinical trial after agreement from the sponsors of the studies concerned (only in the absence of blinding).
* Having agreed to participate in this study by signing the biocollection consent.

Healthy subjects :

* Adult
* Affiliated or beneficiaries of a social security or similar scheme
* Who have agreed to participate in this study by signing the Biocollection consent form.
* No known infectious pathology
* No known history of cancer
* No known history of chronic autoimmune disease
* No background immuno-suppressive treatment

Ancillary Study :

-Metastatic NSCLC with a KRAS G12C mutation, receiving treatment with Sotorasib, Adagrasib, or another KRAS G12C inhibitor, either as monotherapy or in combination.

Exclusion Criteria:

Patients :

* Previous anticancer treatment for Lung cancer
* Patients who have not consented to participate in the BREATHE collection
* History of cancer (excluding thoracic cancer) with evidence of disease for less than 2 years
* Inclusion in a therapeutic trial with blinded treatment
* Patients under guardianship
* Patients with AME.
* Pregnant or breast-feeding women

Healthy subjects :

* Person under guardianship
* Person benefiting from AME (State medical aid)
* Pregnant or breast-feeding women

Ancillary Study :

- Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 5 years
  Overall survival will be defined as the time elapsed between the date of the initial diagnosis of lung cancer and the date of death, regardless of the cause. Patients still alive at the end of the follow-up period will complete their participation in the cohort.

SECONDARY OUTCOMES:
Describe the care pathway for patients with lung cancer. Assess the time intervals between different steps in the initial management of lung cancer. | up to 5 years
  The care pathway will be described through the collection of dates (surgery, radiotherapy, presentation at multidisciplinary consultation meetings, etc.) and types of medical consultations.
Evaluate the return to work for patients of working age who have been treated for lung cancer. | up to 5 years
  Proportion of patients who returned to work after treatment, measurement of the average time taken, and factors associated with the return to work.
Identify specific biomarkers of lung cancer cells (primary tumors or metastatic tissues) in comparison to healthy lung tissues. | up to 5 years
  Quantitative comparison and characterization of biomarkers (extracellular vesicles and miRNA signatures) between tumor tissues and non-cancerous tissues.
Evaluate the prognostic and predictive value of circulating biomarkers at diagnosis and during systemic treatments. | up to 5 years
  Association between levels of circulating biomarkers and overall survival as well as treatment response.

OTHER OUTCOMES:
Predicting the mechanisms of resistance development to KRAS G12C inhibitors through longitudinal analysis of tumor and plasma samples. | up to 5 years
Determining the mechanisms of resistance development to KRAS G12C inhibitors through longitudinal analysis of tumor and plasma samples. | up to 5 years
Determining whether transcriptional changes under sotorasib or adagrasib can predict progression-free survival in patients with metastatic KRAS G12C-mutated NSCLC. | up to 5 years
Assessing the prognostic value of detecting specific molecular alterations occurring under treatment. | up to 5 years
Identifying whether new molecular alterations can be detected in tumor and plasma samples from patients at progression. | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided